CLINICAL TRIAL: NCT01349998
Title: An Open-Label Study to Evaluate the Safety of Long-Term Administration of Product 33525 in Subjects With Tinea Pedis, Tinea Corporis, or Tinea Cruris
Brief Title: Safety of a Topical Antifungal Treatment for Tinea Cruris, Tinea Pedis and Tinea Corporis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tinea Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: MP-1005
Record Dates: First submitted 2011-05-03; First posted 2011-05-09 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Tinea Pedis; Tinea Cruris; Tinea Corporis
MeSH Terms: conditions — Tinea Pedis; Tinea Cruris; Tinea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Safety Population (Experimental)
  Interventions: Drug: Product 33525

INTERVENTIONS:
Drug: Product 33525 — Daily dosing for 2 weeks each recurrence for patients with tinea pedis and Daily dosing for 1 week each recurrence for patients with tinea cruris and tinea corporis

SUMMARY:
The purpose of this study is to examine the long-term safety of treating recurrent episodes of tinea pedis for 14 days for each recurrence and recurrent episodes of tinea corporis or tinea cruris for 7 days for each recurrence with Product 33525.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of tinea cruris, tinea pedis, or tinea corporis. Additional criteria listed in protocol

Exclusion Criteria:

* Pregnancy and allergies. Additional criteria listed in protocol

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Adverse Events | One Year
  To examine the long-term safety of treating tinea pedis, tinea corporis or tinea cruris, treatment-emergent adverse events occurring during the study will be recorded. Adverse events will be summarized by the number of subjects reporting events, system organ class, preferred term, severity, relationship to study drug, and seriousness. Baseline and end of study laboratory assessments will be conducted.

SECONDARY OUTCOMES:
Clinical Cure and Mycological Cure | 1 week Post Treatment, 2 weeks Post Treatment, and 3 weeks Post Treatment
  Proportion of patients achieving effective treatment

CONTACTS AND LOCATIONS:
Locations (24):
- United States (20):
  - Fremont, California
  - Los Angeles, California
  - Miami, Florida
  - Miramar, Florida
  - St. Petersburg, Florida
  - Augusta, Georgia
  - Evansville, Indiana
  - Warren, Michigan
  - Omaha, Nebraska
  - Paramus, New Jersey
  - Albuquerque, New Mexico
  - Cincinnati, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Goodletsville, Tennessee
  - Austin, Texas
  - College Station, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Lynchburg, Virginia
- Belize City, Belize District, Belize
- San Salvador, El Salvador
- San Pedro, Sula, Honduras
- Cidra, Puerto Rico